CLINICAL TRIAL: NCT06611579
Title: A Clinical Study of the inQB8 Transcatheter Tricuspid Valve Replacement System
Brief Title: Clinical Study of the inQB8 TTVR System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: inQB8 Medical Technologies, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-21001
Record Dates: First submitted 2024-09-19; First posted 2024-09-25 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-07

CONDITIONS: Tricuspid Valve Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment (Experimental): Treatment with the inQB8 MonarQ Transcatheter Tricuspid Valve Replacement System
  Interventions: Device: Transcatheter Tricuspid Valve Replacement

INTERVENTIONS:
Device: Transcatheter Tricuspid Valve Replacement — Replacement of the tricuspid valve using a transcatheter approach
  Other Names: inQB8 MonarQ Transcatheter Tricuspid Valve Replacement System

SUMMARY:
Prospective, multi-center study to assess safety and performance of the inQB8 MonarQ Tricuspid Valve Replacement System.

DETAILED DESCRIPTION:
The study is a multi-center, prospective, single-arm study to assess safety and performance of the inQB8 Medical Technologies MonarQ Tricuspid Valve Replacement System.

ELIGIBILITY:
Inclusion Criteria:

* Anatomically suitable for the MonarQ TTVR System
* Symptomatic, tricuspid regurgitation (TR) that is severe or greater
* Adequately treated for heart failure based upon medical standards
* Hemodynamically stable

Exclusion Criteria:

* Need for emergent or urgent surgery for any reason, any planned cardiac surgery within the next 12 months (365 days), or any planned percutaneous cardiac procedure within the next 90 days
* Refractory Heart Failure (HF) that requires or required advanced intervention
* Any condition, in the opinion of the investigator, making it unlikely the patient will be able to complete all protocol procedures and follow-up.
* Currently participating in another investigational biologic, drug or device study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
Absence of device or procedure related major adverse events | 30 days
Change in TR grade from baseline | 30 days

SECONDARY OUTCOMES:
Device and procedure related complications | 30 days and 12 months
  Rate of Device and procedure related complications
NYHA functional classification | 30 days, 6 months, 1 year, and through study completion, an average of 1 year
  Change in NYHA functional class from baseline
Six-minute-walk test | 30 days, 6 months, 1 year, and through study completion, an average of 1 year
  Change in distance from baseline
Health status - KCCQ | 30 days, 6 months, 1 year, and through study completion, an average of 1 year
  Change in quality of life from baseline
TR grade | 30 days, 6 months, 1 year, and through study completion, an average of 1 year
  Change in TR Grade from baseline
Hospitalization | 30 days, 6 months, 1 year, and through study completion, an average of 1 year
  Rate of all-cause hospitalization

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Los Robles Hosptial and Medical Center, Thousand Oaks, California
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - North Shore University Hospital, Manhasset, New York
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Baylor Heart Hospital, Plano, Texas

IPD SHARING:
Plan to Share IPD: No